CLINICAL TRIAL: NCT01673295
Title: RING - Rituximab for Lupus Nephritis With Remission as a Goal, an Investigator-initiated Randomized International Open Multicentric Study
Brief Title: RING - Rituximab for Lupus Nephritis With Remission as a Goal
Acronym: RING
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Frédéric A. Houssiau, MD, PhD (Other)
Responsible Party: Sponsor-Investigator, Frédéric A. Houssiau, MD, PhD, Professeur Ordinaire, Chef de Service Clinique, Université Catholique de Louvain
Organization: Université Catholique de Louvain (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P1200_11
Record Dates: First submitted 2012-08-22; First posted 2012-08-27 (Estimated); Last update posted 2015-05-28 (Estimated); Status verified 2015-05

CONDITIONS: Lupus Nephritis
Keywords: Lupus Nephritis; Rituximab
MeSH Terms: conditions — Lupus Nephritis | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- RTX group (Experimental): Subjects will receive a RTX infusion (1g) at w0, w2, w24, w48 and w72.
  Interventions: Drug: RTX infusions
- Control group (Active Comparator): Subjects will not receive RTX infusions and will be followed in standard of care
  Interventions: Other: Standard of Care

INTERVENTIONS:
Drug: RTX infusions — RTX + Standard of Care
  Arms: RTX group
Other: Standard of Care — Standard of Care only
  Arms: Control group

SUMMARY:
OBJECTIVE To test whether Rituximab (RTX) is efficacious to achieve complete renal response (CR) in Lupus Nephritis (LN) patients with persistent proteinuria (≥1g/d) despite at least 6 months of standard of care (SOC).

STUDY DESIGN Investigator-initiated randomized international open multicentric 104-week study.

DETAILED DESCRIPTION:
After screening (week -8), patients enter in a run-in period of 6 weeks during which treatment is unchanged. At week -2, if persistent proteinuria is confirmed (uP/C ratio ≥1 expressed in mg/mg), patients will be randomized in a 1/1 ratio to 1 of 2 treatment groups as follows :

RTX group Subjects will receive a RTX infusion (1g) at w0, w2, w24, w48 and w72.Control group Subjects will not receive RTX infusions. In both arms, azathioprine (AZA) or mycophenolate mofetil (MMF) will be continued. If prescribed, prednisolone dose should not be > 10 mg/day.

ELIGIBILITY:
Inclusion Criteria:

All the following inclusion criteria are to be met :

1. SLE, according to ACR and/or SLICC (Arthritis Rheum 2012; May 2; doi: 10.1002/art.34473) criteria ;
2. Age ≥15y (except if local ethics committee imposes ≥18y) ;
3. ISN/RPS 2003 Class III (A or A/C), IV (A or A/C ; S or G) or V lupus GN confirmed on renal biopsy performed within 24 months before screening ;
4. Having received one out of four following immunosuppressive regimens:

   i): Euro-Lupus (EL) intravenous (IV) cyclophosphamide (CY) (6x 500 mg q2w) followed by AZA/MMF for 3 months ; ii): NIH IVCY for 6M (6 monthly pulses) followed by AZA/MMF for 3 months ; iii): MMF for at least 6 months at a dose of 2g/day (or the maximal tolerated dose; iv): AZA for at least 6 months at a dose of 2 mg/kg/day (or the maximal toerated dose).

   All patients should be on AZA or MMF at screening. In all regimens, MMF can be replaced by enteric-coated mycophenolic acid (eMPA) ;
5. If on GC, being on maximum 10 mg equivalent prednisolone/d at screening (for at least 2 weeks) ;
6. uP/C ratio ≥1 (expressed in mg/mg) measured in a 24-h urine collection, confirmed at randomization (w-2) ;
7. Contraception (any type ; sexual abstinence is an alternative to contraception in paediatric patients) ;
8. Signed informed consent (drafted according to local practice and approved by the local ethics committee).

Exclusion Criteria:

Any of the following :

1. Recent or ongoing renal flare defined as either i) : fall in estimated glomerular filtration rate (eGFR ; MDRD) ≥25% within 3 month prior to screening or between screening and randomization ; or ii) : increase in urine protein by ≥100% to >3.5g/d compared to previous assessment ;
2. 24-h proteinuria decline >50% over previous 6 months ;
3. Treatment with ≥10 mg equivalent prednisolone/d in the last 2 weeks before screening ;
4. Pregnancy or breast-feeding ;
5. Anticipated non-compliance with the protocol ;
6. History of malignancy (except non-melanoma skin and cervical intraepithelial cancer) ;
7. Previous treatment with RTX (whenever) and previous treatment with another biologic agent within the last 6 months ;
8. HIV infection ;
9. Active HBV/HCV/TB infection ;
10. Severe liver, cardiac, vascular, pulmonary, gastrointestinal, endocrine, neurologic, haematologic or psychiatric disturbances, that would contraindicate inclusion in the protocol, as judged by the clinician.

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 194 (Estimated)
Dates: Start 2014-11; Primary Completion 2015-11 (Estimated); Study Completion 2016-11 (Estimated)

PRIMARY OUTCOMES:
The primary endpoint is the percentage of patients achieving renal complete response (CR) at w104. | 104 weeks
  CR is defined as :
  * uP/C ratio ≤0.5 (expressed in mg/mg) measured in a 24-h urine collection; and
  * eGFR >=60ml/min or, if <60ml/min at screening, not fallen by >20% compared to screening; and
  * no increase of glucocorticoïds (GC) throughout the study (except for two limited courses as per protocol; vide infra); and
  * no introduction of another immunosuppressant.

CONTACTS AND LOCATIONS:
Overall Officials: Frédéric A Houssiau, MD PHD, Principal Investigator — Cliniques universitaires Saint-Luc- Université Catholique de Louvain
Locations (1):
- Cliniques Universitaires Saint Luc, Brussels, Belgium